CLINICAL TRIAL: NCT00165802
Title: A Phase I Open Label Study of E7974 Administered on Day 1 of a 21-Day Cycle In Patients With Advanced Solid Tumors
Brief Title: A Phase I Open Label Study of E7974 Administered on a Day 1 of 21-Day Cycle In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Eisai Medical Services, Eisai Medical Research Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7974-A001-103
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2009-08

CONDITIONS: Cancer, Malignant Tumors
Keywords: Cancer; malignant tumors
MeSH Terms: conditions — Neoplasms | interventions — E 7974

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E7974

INTERVENTIONS:
Drug: E7974 — Maximum Tolerated Dose defined as 0.45 mg/m^2 administered on Day 1 only of a 21-day cycle; the E7974 compound is administered as a bolus infusion; no placebo is given.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of E7974 after bolus IV administration, on Day 1 of a 21-day cycle, to patients with advanced solid tumors that have progressed following effective therapy or for which no effective therapy exists.

DETAILED DESCRIPTION:
The MTD for the Day 1 21-Day schedule was defined at the 0.45 mg/m2 dose level. The study was terminated prior to full enrollment of the colorectal cancer (CRC) expansion cohort, due to a lack of demonstrated activity resulting in Principal Investigator (PI) loss interest to continue enrollment. Collection of all outstanding data is ongoing and database lock is estimated to be complete in June 2008.

ELIGIBILITY:
Inclusion Criteria: At this time, we are only enrolling patients for the MTD cohort that meet all study entry criteria, plus the CRC criterion (Inclusion Criterion #12).Patients who meet all of the inclusion criteria and none of the exclusion criteria will be eligible for entry into the study. Patients must:

1. Have a histologically or cytologically confirmed advanced solid tumor that has progressed following effective therapy or for which no effective therapy exists (including surgery or radiation therapy).
2. Be >= 18 years of age.
3. Have an Eastern Cooperative Oncology Group (ECOG) status of 0, 1, or 2.
4. Have a life expectancy of >= 3 months.
5. Have adequate renal function as evidenced by serum creatinine <= 1.5 mg/dL or creatinine clearance >= 40 mL/minute.
6. Have adequate bone marrow function as evidenced by absolute neutrophil count >= 1,500/µL, hemoglobin of >= 9 g/dL (may be transfused), and platelet count (not transfused) >= 100,000/µL.
7. Have adequate liver function as evidenced by bilirubin <= 1.5 x ULN and alanine transaminase (ALT) and aspartate transaminase (AST) <= 3 times the upper limits of normal (ULN), unless related to liver involvement by tumor, in which case <= 5.0 x ULN.
8. Give written informed consent.
9. Be willing and able to comply with the study protocol for the duration of the study.
10. Be willing to undergo blood draw and urine sampling for PK in Cycle 1.
11. Can have either measurable or non-measurable disease.
12. If a CRC patient is being treated at the MTD, they must have <= 4 prior regimens in the metastatic setting.

Exclusion Criteria:The presence of one or more of the following criteria will disqualify a patient from enrollment in the study:

1. Patients who have received chemotherapy within 3 weeks of E7974 treatment start; (six weeks for nitrosoureas).
2. Patients who have not recovered from any chemotherapy-related or other therapy-related toxicity to < Grade 1 at study entry (excluding alopecia Grade 2).
3. Patients who have received radiotherapy <= 3 weeks prior to study enrollment, (prior radiation therapy allowed to <25% of the bone marrow), and who have not recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia). Lesions that have been radiated cannot be included as sites of measurable disease unless clear tumor progression has been documented in these lesions since the end of radiation therapy.
4. Patients who have had major surgery without full recovery or major surgery within three weeks of E7974 treatment start.
5. Patients with primary brain tumors or metastasis at study entry must have them controlled for > one month by previous treatment, including radiation therapy and /or corticosteroids.
6. Women who are pregnant or breastfeeding.
7. Women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test.
8. Women of childbearing potential unless (1) surgically sterile or (2) physiologically postmenopausal for > 12 months, or (3) using adequate measures (including barrier methods) of contraception.
9. Fertile men or their partners who are not willing to use contraception.
10. Patients who have a history of positive testing for Human Immunodeficiency Virus (HIV) and/or have active hepatitis B or active hepatitis C at study entry.
11. Patients with severe, uncontrolled intercurrent illness or infection.
12. Patients with medically uncontrolled cardiovascular illness defined as unstable angina or congestive heart failure (CHF), with > symptomatic Grade II New York Heart Association (NYHA) Classification, or myocardial infarction (MI) within six months prior to study entry.
13. Patients who have received organ allografts requiring immunosuppressive therapy.
14. Patients who have received investigational drugs including immunotherapy, gene therapy, hormone therapy, biologic therapy, or chemotherapy within the three-week period prior to E7974 treatment start; patients must have recovered from any previous major therapy related toxicity (Grade 3 or 4) to <= Grade 1 at study entry.
15. Patients with a current history of peripheral neuropathy > CTC Grade 2 (e.g., diabetic or chemotherapy-induced neuropathy).
16. Patients with a history of uncontrolled seizures.
17. Patients with other significant diseases or disorders that, in the investigator's opinion, would exclude them from the study.
18. Patients with marked screening or baseline prolongation QT/QTc interval (QTc interval > 470 mm) using the Fridericia method as the main method of QTc analysis.
19. Patients with allergy or hypersensitivity to hemiasterlin based product or analogue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of E7974 in patients with Advanced Solid Tumors. | Duration of each cycle will be 21 days; patients will attend a follow-up visit 30 days after last study treatment. Follow-up for safety and efficacy will occur 6 months after the last patient is accrued to the study.

SECONDARY OUTCOMES:
Assess E7974 for safety, pharmacokinetics (PK) and pharmacodynamics (PD) which will correlate AUC with clinical toxicity and efficacy. | Duration of each cycle will be 21 days; patients will attend a follow-up visit 30 days after last study treatment. Follow-up for safety and efficacy will occur 6 months after the last patient is accrued to the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Zhang, Study Director — Eisai Inc.
Locations (2):
- United States (2):
  - Sylvester Comprehensive Cancer Center - University of Miami, Miami, Florida
  - Cancer Institute Of New Jersey, New Brunswick, New Jersey